CLINICAL TRIAL: NCT05710380
Title: Magnetic Resonance Imaging (MRI) Derived Quantitative Risk Maps for Prostate Cancer Diagnosis Using Targeted Biopsy
Brief Title: MRI Risk Maps for Prostate Cancer Diagnosis Using Targeted Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB22-1311
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Neoplasm
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Single Arm) (Experimental): All participants in this trial will be provided with routine instructions and precaution information before starting the magnetic resonance (MRI) scan. After the MRI, participants will undergo an MRI-guided fusion biopsy of the prostate as ordered by their doctor. During this prostate MRI-guided fusion biopsy, the research team will obtain tissue from up to two additional biopsy targets selected by the Risk Map DSS tool. Ultimately, the clinical radiologist will make the final decision on the targets to be biopsied.
  Interventions: Other: Risk Map Decision Support System (DSS).; Radiation: Magnetic Resonance Imaging (MRI); Procedure: Magnetic Resonance Imaging (MRI) Guided Biopsy

INTERVENTIONS:
Other: Risk Map Decision Support System (DSS). — The Risk Map DSS tool is an image analysis software that automatically interprets images of the prostate that were captured using an MR (magnetic resonance) scanner (an imaging technique that uses scanners to take pictures of the body). This tool can potentially identify additional areas of cancer in your prostate that may have otherwise been missed.
Radiation: Magnetic Resonance Imaging (MRI) — A medical imaging test that uses a large machine/scanner to take images of the body and internal organs and structures.
Procedure: Magnetic Resonance Imaging (MRI) Guided Biopsy — A removal of tumor tissue from the body based on images of the prostate provided by a previous magnetic resonance imaging (MRI) test. Up to 2 biopsies on trial.

SUMMARY:
Doctors leading this study hope to learn about a software that researchers at the University of Chicago have developed to help analyze radiographic images (different techniques for taking images that allow doctors to visualize the body's internal structures) of the prostate. Participation in this research will last about 12 months. There is a one-time MRI and 1-2 biopsies and then the investigator would like to follow the participant's progress.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected prostate cancer who have been referred for a diagnostic magnetic resonance imaging (MRI) exam of the prostate, to be followed by an MRI-guided fusion biopsy of the prostate.
* Voluntary written informed consent before the MRI examination.

Exclusion Criteria:

* Subjects incapable of giving informed written consent.
* Subjects who cannot adhere to the experimental protocols for any reason, or have an inability to communicate with the researcher;
* Subjects with psychiatric disorders that affect their ability to consent for themselves will be excluded and not the entire population of patients with psychiatric disorders.
* Prisoners.
* Minor children (under the age of 18 years old).
* Patients with previous treatments (surgery, radiation, focal ablation, hormone or other chemotherapy) for prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Decision Map Tool Compared to Oncologists | 1 year
  Compare the accuracy of the Risk Map Decision Support Systems (DSS) tool against the clinical accuracy of experienced radiologists in the context of the reference standard of biopsy histology.

CONTACTS AND LOCATIONS:
Overall Officials: Aytekin Oto, MD, Study Chair — University of Chicago Medicine Comprehensive Cancer Center
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF